CLINICAL TRIAL: NCT02428361
Title: Fecal Microbiota Transplant (FMT) for Pouchitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Najwa Elnachef (Other)
Responsible Party: Sponsor-Investigator, Najwa Elnachef, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-15859
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pouchitis patients receiving FMT (Experimental): Pouchitis patients receiving biologically active human fecal material sourced from OpenBiome.The physician will administer 250 mL of the fecal suspension in aliquots of 50-60 mL through the endoscope. The material will be delivered to the most proximal point of insertion.
  Interventions: Drug: Biologically active human fecal material, OpenBiome

INTERVENTIONS:
Drug: Biologically active human fecal material, OpenBiome — Fecal microbiota transplant

SUMMARY:
This is a prospective, open label pilot study in which patients with symptoms of acute or chronic pouchitis will receive FMT therapy delivered via pouchoscopy. The investigators hypothesize that FMT is a safe and effective treatment for patients with pouchitis. Our aims our:

1. To determine if symptoms of pouchitis can be successfully treated by Fecal Microbial Transplantation.
2. To determine if endoscopic appearance of ileal pouch improves following treatment by Fecal Microbial Transplantation.

DETAILED DESCRIPTION:
This is a prospective, open label pilot study in which patients with symptoms of acute or chronic pouchitis will receive FMT therapy delivered via pouchoscopy.

Number of Subjects:

This study will aim to enroll approximately 30 patients with pouchitis.

Eligibility Criteria for FMT Group:

Both acute and chronic pouchitis will be eligible for treatment with FMT. Patients eligible for FMT will include:

1. Patients with history of proctocolectomy with Ileal Pouch-Anal Anastomosis (IPAA) (with pouchitis confirmed by endoscopy and pathology.
2. Concurrent therapies with mesalamine, immunomodulators, corticosteroids and biologic agents will be allowed to continue during study.

All patients who have a pouch for Inflammatory Bowel Disease (IBD) will be evaluated in Gastroenterology clinic or Colorectal surgery clinic. Patients who are eligible for the study will be identified during these regularly scheduled clinic visits. Patients who express interest will be set up for a meeting with a clinical research coordinator who will go over the study in detail and will obtain informed consent.

Prior to the FMT procedure stool samples will be checked for ova and parasites, C. difficile toxin and fecal calprotectin. Serum tests will include erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), Anti-nuclear antibodies (ANA), complete blood cell count, HIV, screening for Hepatitis A, B, C (hep A IgM, hep B surface antigen and antibody, Hep C antibody), and creatinine. Eight days before treatment, patients will take a 5 day course of rifaximin that is discontinued 3 days before FMT treatment.

All patients with clinical suspicion for pouchitis will undergo pouchoscopy. Pouchoscopy (endoscopic evaluation of the pouch) is considered part of standard of care for management of these patients. All participants will undergo a pouchoscopy and this will not be considered a study procedure. This will be done in the endoscopic units at Mt. Zion, Parnassus and/or Mission Bay. During this procedure, for patients in the FMT group, the fecal transplant will take place. For FMT, 250 cc of FMT material (previously screened stool from OpenBiome) will be administered via the endoscope. During each FMT procedure 3 pouch biopsies will be collected. The scope will then be withdrawn and the patient will recover in the endoscopy unit as per protocol.

All patients who have undergone FMT for pouchitis will be called the next day to ensure no adverse events have occurred. A second FMT treatment and a follow up visit will be scheduled 4 weeks after the initial procedure. A pouchoscopy with 3 pouch biopsies will be conducted 6 six months after the initial FMT treatment to check for healing.

One week after the second FMT treatment, patients will be given the option to enroll in a 6 week, once per week FMT capsule therapy to be administered at a 1 hour clinic visit. Patients who receive capsules will be called the following to to ensure no adverse events have occurred.

Study participants will be asked to submit a stool sample prior to treatment, one month after treatment and then after that every three months after treatment up to 1 year in duration for a total of 6 samples. Additionally, blood serum samples will be collected at baseline and again 1 and 6 months after FMT procedure. Study participants will also be administered a patient survey to assess their clinical outcomes/symptoms prior to treatment and again 1 month after receiving treatment. In addition, all patients will receive a phone call 24 hours, 1 week, 1 month and and then every 3 months for 3 years after FMT treatment.

ELIGIBILITY:
Inclusion Criteria:

Both acute and chronic pouchitis will be eligible for treatment with FMT. Patients eligible for FMT will include:

1. Patients with history of proctocolectomy with IPAA with pouchitis confirmed by endoscopy and pathology.
2. Concurrent therapies with mesalamine, immunomodulators, corticosteroids and biologic agents will be allowed to continue during study.

Exclusion Criteria:

1. Female patients who are pregnant.
2. Patients with severe immunosuppression (absolute neutrophil count < 1000 or CD4 count <200).
3. Patients with diagnosis of ileal Crohn's Disease.
4. Patients with untreated enteric infection.
5. Patients with fistulizing disease.
6. Patients with gastroparesis or dysphagia will not be eligible for the arm of the study allowing for administration of weekly capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of pouchitis | 4 weeks
  In order to assess clinical improvement of pouchitis, patients will be scheduled for a 4 week post-FMT treatment clinic visit to ensure no adverse events have occurred and to assess patient symptoms.
  Patients will also complete a survey both before and after treatment to evaluate the efficacy of FMT treatment.

SECONDARY OUTCOMES:
Mucosal healing | 6 months
  repeat pouchoscopy to determine

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Division of Gastroenterology at Mount Zion, San Francisco, California, United States